CLINICAL TRIAL: NCT03302143
Title: A Comparative, Randomized, Prospective, Clinical Study to Evaluate the Facial Bone and Esthetic Outcome of Buccal Augmentation Bone Grafting Techniques in Early (Type 2) Implant Placement
Brief Title: Radiographic and the Esthetic Outcome of Two Different Bone Grafting Techniques in Early Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC20120264H
Record Dates: First submitted 2017-09-26; First posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Missing Tooth; Fractured Tooth
Keywords: Dental Implant; Guided Bone Regeneration; Contour Augmentation
MeSH Terms: conditions — Anodontia; Tooth Fractures

STUDY DESIGN:
Intervention Model Description: A comparative, randomized, prospective, clinical study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): Guided bone regeneration with Bovine Bone Mineral
  Interventions: Procedure: Guided bone regeneration with Bovine Bone Mineral
- Experimental (Experimental): Guided bone regeneration with freeze dried bone allograft
  Interventions: Procedure: Guided bone regeneration with freeze dried bone allograft

INTERVENTIONS:
Procedure: Guided bone regeneration with Bovine Bone Mineral — Guided bone regeneration with Bovine Bone Mineral
  Arms: Control
Procedure: Guided bone regeneration with freeze dried bone allograft — Guided bone regeneration with freeze dried bone allograft
  Arms: Experimental

SUMMARY:
Total of 48 subjects were randomly assigned to treatment groups:

UT Health Science Center at San Antonio Chi Mei Medical Center, Tainan, Taiwan

Patients require a maxillary non-molar extraction site that is planned to be replaced by a dental implant and crown. This includes Straumann BL SLActive: Narrow (3.3mm) & Regular (4.1mm) Crossfit implants in all available lengths.

Patients were randomly selected to receive either FDBA (test) or Autogenous bone + DBBM (control/standard) for contour augmentation.

DETAILED DESCRIPTION:
This comparative, randomized, prospective clinical study is designed to compare clinical outcomes and facial bone height and thickness of two different bone grafting techniques after augmentation in (Type 2) early implant placement.

Human subjects who could potentially qualify with the said inclusion criteria will be evaluated and screened. 24 human subjects who qualify for the procedure will have a thorough evaluation performed after obtaining consent from the patient. All subjects will require extraction of maxillary teeth (incisors, canines, premolars), followed by early implant placement of the missing teeth after 4 to 8 weeks extraction.

There will be two subject groups in this study in which the 24 human subjects in will randomly be placed by selecting the number "1" or "2" from a hat. 24 human subjects will be divided into two groups including 12 subjects using control group design and 12 subjects using test group design. 12 subjects will be placed randomly into Group 1 and will undergo the flapless extraction and early implant placement with GBR procedure using the control group design. 12 subjects will be placed randomly into Group 2 and will undergo the flapless extraction and early implant placement with GBR procedure using the test group design.

During the implant placement visit after 4 to 8 weeks of extraction, patient will be asked to select a number from a hat. If the number showed "1" as a control group, autograft , BBM and collagen membrane will be used as GBR materials after implant placement. If the number showed "2" as a test group, FDBA and collagen membrane will be used as GBR materials after implant placement.

Extraction sites will include maxillary teeth (11,12,13,14,15,21,22,23,24,25 according to FDI) having intact adjacent teeth. Implants placed for this study will have a SLActive surface, bone level design, Straumann NC 3.3mm or RC 4.1mm in diameter at all available implant lengths.

Control group: early implant placement with autograft plus BBM (Bio-Oss, Geistlich Pharm AG, Wolhausen, Switzerland) plus two layers of collagen membrane (BioGide®).

Test group: early implant placement with FDBA (Straumann Allograft GC®) plus two layers of collagen membrane (BioGide®).

These procedures will follow the guidelines as described by Buser et al. (2008). Implant placements will follow standard protocols utilizing tapping and placement with the hand ratchet.

A CBCT radiograph will be made during the screening visit to determine eligibility for the study and immediately following implant placement with GBR procedure to provide facial bone height and thickness measurements. The second CBCT procedure is not typically a standard of care procedure. After 12 months post loading healing time, the patient will receive another CBCT. This CBCT is also not a standard of care procedure but can accurately assess the amount of facial bone height and thickness maintained during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is 18 years or older.
2. Non-smoker or patient has smoking habit and < 1 pack per day.
3. Ability to understand and provide informed consent before starting the study.
4. Ability and willingness to comply with all study requirements.
5. The patient, if of child-bearing potential, has a negative urine pregnancy test.
6. Adequate oral hygiene to allow for implant therapy consistent with standards of care.
7. Adequate primary stability following early implant placement protocols utilizing Straumann Bone Level implants NC 3.3mm or RC 4.1mm in diameter at all available implant lengths.
8. One or more teeth in maxilla (11,12,13,14,15,21,22,23,24,25 according to FDI) has been identified as having a hopeless prognosis requiring extraction leading to a single-tooth gap requiring implant placement as determined by clinician.
9. Implant site that has a defect and requires bone augmentation. This will be determined by measuring on the CBCT image the available space for the implant and whether or not there is enough bone width where the implant is to be placed.

Exclusion Criteria:

1. Patient reports current smoking habit > 1 pack per day or tobacco chewing use.
2. History of alcoholism or drug abuse within the past 5 years.
3. Severe bruxism or clenching habits.
4. Patient has significant untreated periodontal disease (grade III or IV), caries, or clinical or radiographic signs of infection within two adjacent tooth positions of implant area.
5. History of HIV infection, Hepatitis B or C.
6. Patients with a history of systemic disease that precludes standard dental implant therapy.
7. Presence of local inflammation or mucosal diseases such as lichen planus
8. Patient history consistent with high risk for subacute bacterial endocarditis
9. Current hematological disorder or coumadin (or similar) therapy
10. Patient currently undergoing chemotherapy
11. Patient history of radiation treatment to the head or neck
12. Physical or mental handicaps that would interfere with patient's ability to exercise good oral hygiene on a regular basis
13. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-07-30 (Actual); Primary Completion 2016-05-15 (Actual); Study Completion 2016-05-15 (Actual)

PRIMARY OUTCOMES:
Facial bone thickness | Measured at 1 year post-loading
  Facial bone thickness 1 year post-loading at 1, 3, and 5mm from the implant platform

SECONDARY OUTCOMES:
Change in facial bone thickness | Between implant placement and 1 year post-loading
  Change in facial bone thickness between implant placement and 1 year post-loading
mPI measurement | Measured at 6 and 12-months post-loading
  Measurement of modified Plaque Index
PD measurement | Measured at 6 and 12-months post-loading
  Measurement of pocket depth
mSBI measurement | Measured at 6 and 12-months post-loading
  Measurement of modified sulcus bleeding index
KM measurement | Measured at 6 and 12-months post-loading
  Measurement of keratinized mucosa